CLINICAL TRIAL: NCT05742022
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled Clinical Trial of Safety and Efficacy of "Phospholipovit" in Patients With Combined Hyperlipidemia
Brief Title: "Phospholipovit" vs Placebo in Patients With Combined Hyperlipidemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Biomedical Chemistry, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05F
Record Dates: First submitted 2023-02-01; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Combined Hyperlipidemia
Keywords: Phospholipid nanoparticles; non-HDL-C level; TG level

STUDY DESIGN:
Intervention Model Description: At clinical centers, patients will be equally randomized by the "envelope method" into two groups to receive "Phospholipovit" or placebo.
  The drugs will be administered after the signed informed consent. "Phospholipovit" will be administered 500 mg orally 2 times a day, for 12 weeks. Placebo will be administered orally 2 times a day, for 12 weeks. All patients will be examined after 12 weeks.
Who Masked: Participant, Care Provider
Masking Description: two or more parties are unaware of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Phospholipovit" (Experimental): Powder for preparing a solution for oral administration. 500 mg orally 2 times a day, for 12 weeks
  Interventions: Drug: "Phospholipovit"
- Placebo (Experimental): Powder for preparing a solution for oral administration. 500 mg orally 2 times a day, for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: "Phospholipovit" — 500 mg orally 2 times a day, for 12 weeks
  Arms: "Phospholipovit"
Drug: Placebo — 500 mg orally 2 times a day, for 12 weeks
  Arms: Placebo

SUMMARY:
"Phospholipovit" vs placebo in patients with combined hyperlipidemia

DETAILED DESCRIPTION:
It is well known that atherosclerosis and its complications are the leading cause of morbidity and mortality in the world, and the high blood cholesterol is one of the leading risk factors for atherosclerosis.

Among cholesterol-lowering agents, the most common are inhibitors of HMG-CoA reductase, so-called statins. Nevertheless, low attention is paid to the process responsible for cholesterol removing from the cells - the so-called "reverse cholesterol transport" (RCT). The major lipoproteins, involved in RCT, are high-density lipoproteins (HDL). The effectiveness of RCT is determined not only by the level of cholesterol in HDL, but also by the composition of HDL, in particular, by the content of phosphatidylcholine (PC) in HDL.

Based on the original phospholipid composition, the Institute of Biomedical Chemistry developed the "Phospholipovit" - the aqueous medium of nanoemulsion of phospholipids with a particle size of 20-25 nm. The intestinal absorption of phospholipids nanoemulsion should contribute to the HDL enrichment by phospholipids, and, consequently, to the enhancement of RCT. A study of the safety and tolerability of the "Phospholipovit" in healthy patients has been completed. The "Phospholipovit" has demonstrated safety and tolerability.

The main objective of this study is to evaluate the effectiveness and safety of "Phospholipovit", a powder for preparation of an oral solution, 500 mg compared with placebo in patients with combined hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Availability of signed and dated informed consent of the patient to participate in the study;
* Patients with moderate combined hyperlipidemia, defined as:

Total cholesterol level 3 - 7 mmol/l, LDL-C 2.5 - 5 mmol/l, TG 1.7 - 4.5 mmol/l, and HDL-C < 1 mmol/l during screening for men and < 1.2 mmol/l for women;

* Patient consent to use reliable contraceptive methods throughout the study;
* The patient's ability to adequately cooperation.

Exclusion Criteria:

* TG > 4.5 mmol/l;
* Total cholesterol >7 mmol/l;
* LDL cholesterol >5 mmol/l;
* Age less than 30 or older than 75;
* Diseases or metabolic disorders that can cause an increase in LDL-C, total cholesterol and TG (secondary dyslipidemia);
* Patients receiving high doses of statin drugs (rosuvastatin ≥40 mg, atorvastatin ≥80 mg);
* Any acute or exacerbation of chronic infectious diseases;
* Type 1 Diabetes mellitus;
* Glomerular filtration rate less than 30 ml/min/1.73 m2;
* Patients who have undergone acute conditions (infections, injuries, operations) in the period less than 2 months before the start of the study;
* Patients with severe dysfunction of the liver and/or kidneys, and/or other vital organs, accompanied by decompensation of their functions; diseases of the central nervous system, with severe impairment of cognitive and mnestic functions;
* Persistent increase in liver enzymes activity (transaminases) of unclear etiology or increased liver enzymes activity by 2 or more times from the upper limit of the norm;
* Alcohol abuse more than 5 units of alcohol per week (1 unit alcohol is equivalent to 0.325 liters beer, 130 ml wine, 30 ml alcohol);
* Drug use;
* A history of a positive HIV test result;
* Positive test result for hepatitis B and C, syphilis;
* A history of hypothyroidism or thyroid-stimulating hormone levels (TSH) exceeding > 1X upper limit of normal (ULN) during screening;
* History of oncological disease during the last 5 years;
* Patients diagnosed with porphyria;
* Patients diagnosed with myopathy;
* Clinically significant abnormal blood test results general urinalysis at screening;
* Hypersensitivity to phospholipids or any components of investigational drug;
* Indications for drug therapy a list of therapies prohibited during the study;
* Any other diseases or conditions that, in the opinion of the investigator, may distort the results of the study and limit the patient's participation in the study;
* Pregnancy and lactation;
* Patient participation in another clinical trial or use of any investigational drug during 1 month prior to inclusion in the study;
* Not using contraception for patients of reproductive age.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in non-HDL-C values | week 12
  The efficacy is evaluated in terms of the percentage change from baseline in non-HDL-C values

SECONDARY OUTCOMES:
Dynamics of change of total cholesterol level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of total cholesterol level compared with the baseline
Dynamics of change of LDL-C level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of LDL-C level compared with the baseline
Dynamics of change of HDL-C level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of HDL-C level compared with the baseline
Dynamics of change of TG level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of TG level compared with the baseline
Dynamics of change of VLDL-C level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of VLDL-C level compared with the baseline
Dynamics of change of Apo-A1 level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of Apo-A1 level compared with the baseline
Dynamics of change of Apo-B level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of Apo-B level compared with the baseline
Dynamics of change of LP (a) level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of LP (a) level compared with the baseline
Dynamics of change of atherogenic index compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of change of atherogenic index compared with the baseline
Dynamics of average hs-CRP level compared with the baseline | week 12
  The efficacy is evaluated in terms of the dynamics of average hs-CRP level compared with the baseline
Change in composition and particle size of fasting HDL-C, LDL-C and VLDL-C compared with the baseline | week 12
  The efficacy is evaluated in terms of the change in composition and particle size of fasting HDL-C, LDL-C and VLDL-C compared with the baseline (limited sample of patients)

OTHER OUTCOMES:
Safety endpoint - Number and severity of serious adverse events (SAEs) and AEs in organs and systems | within 12 weeks
  The safety is evaluated in terms of the number and severity of SAEs and AEs in organs and systems
Safety endpoint - The frequency of cases of early termination of participation in the study due to the development AE and SAE | within 12 weeks
  The safety is evaluated in terms of the frequency of cases of early termination of participation in the study due to the development AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Alexander I. Archakov, MD, PhD, Principal Investigator — Institute of Biomedical Chemistry
Locations (3):
- Russia (3):
  - Federal State Budgetary Institution "National Medical Research Centre Of Cardiology" of the Ministry of Health of the Russian Federation, Moscow
  - LLC "Nizhny Novgorod Medical clinic", Nizhny Novgorod
  - LLC "Medical Center for Diagnostics and prevention plus", Yaroslavl

IPD SHARING:
Plan to Share IPD: No